CLINICAL TRIAL: NCT03447860
Title: Practice of Acceptance, Awareness, and Compassion in Caregiving (PAACC): A Randomized Controlled Trial on the Effectiveness of a Mindfulness Based Caregiver Multicomponent Intervention
Brief Title: Practice of Acceptance, Awareness, and Compassion in Caregiving (PAACC)
Acronym: PAACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salem Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); Virginia Polytechnic Institute and State University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mamta Sapra, Geriatric psychiatrist, MD, Salem Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS0010
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REACH-VA (Active Comparator): A cognitive-behavior based multi-component caregiver intervention to reduce caregiver stress.
  Interventions: Behavioral: REACH-VA
- PAACC (Experimental): A mindfulness-based multi-component caregiver intervention to reduce caregiver stress.
  Interventions: Behavioral: PAACC

INTERVENTIONS:
Behavioral: PAACC — Mindfulness based caregiver intervention that includes education , problem solving, skill building, stress management and mindfulness to help enhance compassion and acceptance of self and others
  Arms: PAACC
Behavioral: REACH-VA — A cognitive-behavior based multi-component caregiver intervention to reduce caregiver stress
  Arms: REACH-VA

SUMMARY:
The Primary objective of the study is to evaluate the effectiveness of mindfulness based caregiver intervention, Practice of Acceptance, Awareness, and Compassion in Caregiving (PAACC) compared to an established cognitive behavior therapy based dementia caregiver intervention, Resources for Enhancing Alzheimer's Caregiver Health (REACH) in improving caregiver burden and quality of life of care recipient.

DETAILED DESCRIPTION:
The study is a randomized controlled trial comparing a mindfulness-enhanced evidence-based caregiver skill-building intervention (PAACC) to REACH-VA to reduce caregiver burden and increase quality of life of the care recipient. For this, caregivers of persons with ADRD or TBI-AD who have moderate to severe burden will be randomly assigned to either receive PAACC or receive REACH-VA. Both the interventions will include 4 biweekly sessions delivered by trained interventionists, followed by an outcome testing session after the intervention. Outcomes of caregiver stress, health and well being will be assessed at baseline and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers will include family members living with the individual diagnosed with Alzheimer's Disease( AD) or Alzheimer's disease related dementia(ADRD) or Traumatic Brain Injury -AD(TBI-AD) with moderate to severe caregiver burden .
* Care recipients with diagnosis of Diagnosis of AD or ADRD or TBI-related AD .

Exclusion Criteria:

* Care givers: Determined to be an imminent risk to self or others,the Care recipient currently resides in a nursing home or assisted living facilities, unable to provide their own consent to participate in the study , and active substance use disorder in the last 1yr.
* Care recipient: Determined to be an imminent risk to self or others, Caregiver is not interested in the study, unable to obtain informed consent from the Care recipient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | 4-6 weeks
  The Perceived Stress Scale (PSS) is a 10-item self-report scale developed to measure the degree to which each participant perceives and appraises recent life events as stressful

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Sapra, MD, Principal Investigator — Salem VAMC
Locations (2):
- United States (2):
  - VA Boston Health Care system, Brockton, Massachusetts
  - Salem VAMC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No